CLINICAL TRIAL: NCT02917629
Title: Phase IIB Randomized, Placebo-Controlled Trial of ACTOplus Met® XR in Subjects With Stage I-IV Squamous Cell Carcinoma of the Oral Cavity or Oropharynx Prior to Definitive Treatment
Brief Title: ACTOplus Met XR in Treating Patients With Stage I-IV Oral Cavity or Oropharynx Cancer Undergoing Definitive Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual combined with expiration of study drug
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2016-01407; NCI-2016-01407 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UW16110; N01-CN-2012-00033; UWI2016-07-01 (Other: University of Wisconsin Hospital and Clinics); UWI2016-07-01 (Other: DCP); N01CN00033 (NIH); P30CA014520 (NIH)
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Oral Cavity Neoplasm; Oropharyngeal Neoplasm; Stage 0 Oral Cavity Squamous Cell Carcinoma American Joint Committee on Cancer (AJCC) v6 and v7; Stage 0 Oropharyngeal Squamous Cell Carcinoma AJCC v6 and v7; Stage I Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage I Oropharyngeal Squamous Cell Carcinoma AJCC v6 and v7; Stage II Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage II Oropharyngeal Squamous Cell Carcinoma AJCC v6 and v7; Stage III Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage III Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVA Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVB Oropharyngeal Squamous Cell Carcinoma AJCC v7
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (ACTOplus met XR) (Experimental): Patients receive ACTOplus met XR PO QD for 10-21 days in the absence of disease progression or unacceptable toxicity. Patients may continue ACTOplus met XR PO QD for a maximum of 25 days if end of treatment biopsy/surgical treatment is delayed beyond day 22.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Metformide Hydrochloride/Pioglitazone Hydrochloride Extended-Release Tablet; Other: Pharmacological Study
- Group II (placebo) (Placebo Comparator): Patients receive placebo PO QD daily for 10-21 days.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Metformide Hydrochloride/Pioglitazone Hydrochloride Extended-Release Tablet — Given PO
  Other Names: ACTOplus Met XR; Metformide HCl/Pioglitazone HCl ER Tablet
  Arms: Group I (ACTOplus met XR)
Other: Pharmacological Study — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group II (placebo)

SUMMARY:
This randomized phase IIb trial studies how well ACTOplus met extended release (XR) works in treating in patients with stage I-IV oral cavity or oropharynx cancer that are undergoing definitive treatment. Chemoprevention is the use of drugs to keep oral cavity or oropharynx cancer from forming or coming back. The use of ACTOplus met XR may slow disease progression in patients with oral cavity or oropharynx cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether 10-21 days of treatment with ACTOplus met XR will result in a decrease in proliferation index (Ki-67) expression in oral cavity/oropharyngeal tumor tissue as compared to placebo.

SECONDARY OBJECTIVES:

I. Compare differences in proliferation index (Ki-67) expression from baseline to post-exposure in visually normal appearing oral cavity/oropharyngeal tissue.

II. Compare immunohistochemical differences in the apoptosis biomarker cleaved caspase 3 from baseline to post-exposure in oral cavity/oropharyngeal adjacent visually normal appearing tissue and tumor tissue samples.

III. Compare immunohistochemical differences from baseline to post-exposure in oral cavity/oropharyngeal tumor tissue samples with regard to cyclin D1, p21 and biguanide or PPAR gamma associated pathway biomarkers; prospective biomarkers on the panel will include phosphorylated (p)AKT, pAMPK, pS6 (metformin), and PPAR gamma.

IV. Compare immunohistochemical differences from baseline to post-exposure of oral cavity/oropharyngeal tumor tissue samples with regard to tumor infiltrating immune cells (effector CD8 [CD8+]), regulatory CD4 T regulatory (Treg) (CD4+Foxp3+), tumor associated myeloid cells (CD68), PD1 and PD-L1.

V. Compare and correlate pre- and post-ACTOplus met XR treatment human ribonucleic acid (RNA)-sequencing (seq) gene analysis on total RNA samples from oral cavity/oropharyngeal adjacent visually normal appearing tissue and tumor tissue pre-and post-study treatment.

VI. Determine human papillomavirus (HPV) status in pre-treatment tumor tissue using p16 immunohistochemistry.

EXPLORATORY OBJECTIVES I. Compare pre- and post-study treatment fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/computed tomography (CT) scans with regard to standardized uptake value (SUV) of FDG and tumor burden using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 in those participants with a preintervention standard of care staging FDG-PET/CT.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive ACTOplus met XR orally (PO) once daily (QD) for 10-21 days in the absence of disease progression or unacceptable toxicity. Patients may continue ACTOplus met XR PO QD for a maximum of 25 days if end of treatment biopsy/surgical treatment is delayed beyond day 22.

GROUP II: Patients receive placebo PO QD daily for 10-21 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a newly diagnosed, histologically confirmed, stage I-IV squamous cell carcinoma or squamous cell carcinoma in situ of the oral cavity or oropharynx and will be undergoing definitive surgical, radiotherapy, or chemoradiation treatment; patients who are NOT candidates for localized treatment (surgery, radiation or chemoradiation) with curative intent (i.e.patients with distant metastasis or contra-indication to localized treatment) are not eligible OR
* Participant has a lesion in the oral cavity or oropharynx that is not yet biopsied but is highly suspicious for cancer; (randomization will be placed on hold until the presence of cancer is histologically confirmed, and a treatment plan is established; if the presence of cancer is not confirmed, the participant will be considered a screen failure)
* The participant's primary tumor is accessible for the collection of 4 mm samples of tumor and adjacent visually normal appearing tissue for biomarker analysis and the participant is willing to have these samples collected at baseline and at the end of study visit. (The protocol requires the collection of fresh tissue for biomarker analysis)

  * Patients who have not yet had a diagnostic biopsy:

    * The tissue samples for biomarker analysis may be collected in conjunction with the patient's standard of care diagnostic biopsy but not until after the patient has signed informed consent and it has been determined that they meet all of the eligibility criteria for this protocol with the exception of normal organ and marrow function as defined by the clinical laboratory test results listed for that criterion. In this situation, because the patient would be having a biopsy regardless of whether or not they were participating in this study, it is not required to obtain these results prior to conducting the biopsy. It is however, required to confirm normal organ and marrow function prior to randomization.
    * Patients who are scheduled for a direct operative laryngoscopy with biopsy (DL biopsy) for diagnostic purposes may be candidates for this study provided the following criteria are met:

      * The lesion to be biopsied is within the anatomic confines of the oropharynx (i.e. above the epiglottis).
      * Tissue samples for biomarker analysis of the required 4 mm size are able to be obtained from both the lesion and an area of visually normal appearing tissue adjacent to but 1 cm distant from the lesion.

In this situation, randomization will be placed on hold until the following criteria are met:

* Normal organ and marrow function is confirmed.
* There is histologic confirmation of squamous cell carcinoma.
* It has been determined that surgical excision will be the first line standard of care treatment and the end of study tissue samples will be obtained in conjunction with that surgery.

Because these patient's lesions are not accessible to end of study tissue sample collection in the outpatient clinic setting, the only way to obtain those samples is in conjunction with standard of care surgical excision of the lesion. If the first line of treatment will be non-surgical, the patient will be considered a screen failure. Under no circumstances will DL biopsy be used for the sole purpose of collecting tissue samples for biomarker analysis.

* Patients who have already had a diagnostic biopsy:

  * The baseline tissue samples for biomarker analysis will be collected in the outpatient clinic setting as a "for research purposes only" procedure. The samples may not be collected until it has been determined that the participant meets all eligibility criteria for this protocol.
* End of study tissue sample collection:

  * If surgical excision will be the patient's first line treatment, the end of study tissue samples for biomarker analysis will be collected in conjunction with that surgery. If, for any reason, the patient's surgery is delayed beyond Day 26, the end of study tissue samples may be collected in the outpatient clinic setting.
  * If the patient's first line of treatment will not be surgical excision, the end of study tissue samples for biomarker analysis will be collected in the outpatient clinic setting prior to initiation of the non-surgical treatment.

    * Participant is able to complete a minimum of 10 days of study agent dosing prior to initiation of definitive treatment for their cancer
    * Participant is scheduled for an end of study biopsy within 22 days of starting study agent and within 52 days of their study screening visit; (if the participant is scheduled for surgical excision of the tumor and the surgery is delayed for any reason after the participant has started taking the study agent, study agent dosing may be extended up to a maximum of 25 days without compromising the evaluability of the end of study biomarkers)
    * Eastern Cooperative Oncology Group (ECOG) performance status = 0 or 1
    * Life expectancy is > 6 months
    * Body mass index (BMI) is >= 18.5
    * Hemoglobin >= 10 g/dl
    * White blood cells >= 3,000/microliter
    * Platelets >= 100,000/microliter
    * Total bilirubin =< 1.2 x institutional upper limit of normal
* With the exception of candidates with a diagnosis of Gilbert's disease in which case the total bilirubin may extend up to 1.5 x institutional upper limit of normal

  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 1.2 x institutional upper limit of normal
  * Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.2 x institutional upper limit of normal
  * Glucose, serum < 200 mg/dL
  * Estimated glomerular filtration rate (eGFR) > 45 mL/min (if eGFR is not included on the clinical lab report, the chronic kidney disease epidemiology [CKD-EPI] creatinine calculator may be used)
  * Participant is able to swallow a tablet whole
  * Participant is willing and able to participate for the duration of the study
  * Participant of childbearing potential agrees to use adequate contraception (a hormonal method that has been in continual use for a minimum of 3 months prior to the study screening visit, a barrier method, or abstinence) for the duration of their study participation. (Therapy with pioglitazone may result in ovulation in some premenopausal anovulatory women. In addition, the effects of ACTOplus Met XR on the developing human fetus at the recommended therapeutic dose are unknown. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.)
* Note: Due to the risks associated with hormonal methods of birth control, participants should not start hormonal therapy for the purpose of meeting the eligibility criteria for this protocol.

  * Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participant has received or will receive some form of treatment for their cancer prior to completing a minimum of 10 days of study agent dosing; (a biopsy is not considered a form of treatment)
* Participant has a concurrent diagnosis of type I or type II diabetes that is being treated with insulin or an oral antidiabetic agent; (participants whose type II diabetes is controlled with diet and/or exercise alone are eligible provided they meet all other eligibility criteria)
* Participant has taken any of the following medications within the past 3 months:

  * A thiazolidinedione (e.g. pioglitazone [Actos] or rosiglitazone [Avandia]),
  * A biguanide (e.g. metformin [Glucophage, Glumetza, Fortamet, Riomet] or proguanil [Paludrine])
  * A combination drug containing one of the agents above (brand names include: ACTOplus Met, Avandamet, Avandaryl, Duetact, Glucovance, Invokamet, Janumet, Jentadueto, Komboglyze, Metaglip, PrandiMet, Synjardy, Xigudo)
* Participant is currently taking a strong CYP2C8 inhibitor (e.g. gemfibrozil [Lopid])
* Participant is currently taking an enzyme inducer of CYP2C8 (carbamazepine [Carbatrol, Epitol, Equetro, Tegretol] cortisol [Hydrocortisone]; dexamethasone [Decadron]; phenobarbital [Luminal Sodium]; phenytoin [Dilantin, Phenytek, Novaplus Phenytoin Sodium]; primidone [Mysoline]; rifampin [Rifadin, Rimactane]; rifapentine [Priftin]; secobarbital [Seconal])
* Participant is currently taking topiramate (Topamax) commonly used in epilepsy or to prevent migraines or other carbonic anhydrase inhibitors (e.g. zonisamide [Zonegran]; acetazolamide [Diamox Sequels]; or dichlorphenamide [Keveyis, Daranide])
* Participant is currently taking a cationic drug or multidrug and toxin extrusion [MATE] inhibitor (e.g. amiloride [Midamor]; cimetidine [Tagamet]; digoxin [Lanoxin, Digitek, Digox]; dolutegravir [Tivicay]; morphine [Roxanol, Duramorph, Kadian, MS Contin]; procainamide [Pronestyl, Procanbid]; quinidine [Quinidex, Cardioquin, Quin-G, Quinora]; quinine [Qualaquin, Quinamm, Quiphile]; ranitidine [Zantac, Deprizine, Gabitidine]; ranolazine [Ranexa]; triamterene [Dyrenium)] trimethoprim [Proloprim, Trimpex, Primsol]; vancomycin [Vancocin, Vancoled]; or vandetanib [Calpresa])
* Participants is taking another investigational agent
* Participant has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ACTOplus Met XR
* Participant has a contraindication to biopsy
* Participants with a history of congestive heart failure or New York Heart Association (NYHA) class III or IV functional status are excluded
* Participant has a history of liver disease
* Participant has > Common Terminology Criteria for Adverse Events (CTCAE) grade 1 limb edema (5 - 10% inter-limb discrepancy in volume or circumference at point of greatest visible difference; swelling or obscuration of anatomic architecture on close inspection)
* Participant has a history of hypoglycemia
* Participant is an active alcoholic or consumes excessive amounts of alcohol per the following definitions:

  * Female: More than 3 drinks on any day or a total of more than seven drinks in a week
  * Male: More than 4 drinks on any day or a total of more than 14 drinks in a week

    * 1 drink =

      * Beer: 12 oz. (1 standard size can or bottle)
      * Wine: 5 oz. (one standard glass)
      * Spirits: 6 oz. (one mixed drink or one 1.5 fluid oz. shot)
* Participant has a history of macular edema
* Participant has a history of bladder cancer (including in situ bladder cancer)
* Participant has a history of invasive cancer (other than non-melanoma skin cancer or cervical cancer in situ) active within 18 months prior to the baseline study visit; (participants who have a history of cancer that was curatively treated without evidence of recurrence in the 18 months prior to the baseline study visit are considered eligible)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Participant is pregnant, breast feeding or planning to become pregnant; (all participants of childbearing potential regardless of method of birth control must have a negative pregnancy test at baseline; a woman is considered not to be of childbearing potential if she has had a hysterectomy, bilateral oophorectomy, or if she is > 55 years of age with >= 2 years of amenorrhea)

  * Breastfeeding should be discontinued if the mother is treated with ACTOplus met XR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank G Ondrey, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Rochester, Rochester, New York
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from Johns Hopkins University - Sidney Kimmel Comprehensive Cancer Center, UW Hospital and Clinics, and University of Minnesota - Masonic Cancer Center between May 31, 2018 and August 2, 2019.
Pre-assignment Details: 16 people were consented and 10 people were subsequently determined to be ineligible. 6 participants were randomized to study.
Groups:
- Group I (ACTOplus Met XR): Patients receive ACTOplus met extended release (XR) by mouth (PO) once a day (QD) for 10-21 days in the absence of disease progression or unacceptable toxicity. Patients may continue ACTOplus met XR PO QD for a maximum of 25 days if end of treatment biopsy/surgical treatment is delayed beyond day 22.
  Laboratory Biomarker Analysis: Correlative studies
  Metformide Hydrochloride/Pioglitazone Hydrochloride Extended-Release Tablet: Given PO
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Group I (ACTOplus Met XR) | Group II (Placebo)
Started | 4 | 2
Considered Study Compliant | 4 | 1
Experienced Study Drug Interruption | 2 | 1
Completed | 4 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (ACTOplus Met XR) | Group II (Placebo) | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) describes a person's function and ability to care for themself. 0 is fully active, 1 is restricted, 2 is capable of self-care but unable to carry out work activities, 3 is capable of limited self-care and confined to bed or chair more than 50% of waking hours, 4 is completely disabled and confined to bed or chair, and 5 is dead.
  Participants
    0 (Fully Active) | 4 | 2 | 6
    1 (Restricted) | 0 | 0 | 0
Systolic Blood Pressure [Mean (Full Range); unit: mmHg] | 141.75 [124 to 155] | 135.00 [131 to 139] | 139.50 [124 to 155]
Diastolic Blood Pressure [Mean (Full Range); unit: mmHg] | 80.00 [68 to 91] | 86.00 [75 to 97] | 82.00 [68 to 97]
Pulse [Mean (Full Range); unit: beats per minute] | 66.00 [59 to 74] | 79.00 [79 to 79] | 70.34 [59 to 79]
Temperature [Mean (Full Range); unit: degrees Fahrenheit (F)] | 97.92 [97.40 to 98.30] | 98.05 [98.00 to 98.10] | 97.96 [97.40 to 98.30]
Height [Mean (Full Range); unit: centimeters] | 171.48 [161.29 to 177.80] | 180.00 [172.01 to 188.00] | 174.32 [161.29 to 188.00]
Weight [Mean (Full Range); unit: kilograms] | 88.64 [73.53 to 101.30] | 93.67 [79.83 to 107.50] | 90.32 [73.53 to 107.50]
Body Mass Index (BMI) [Mean (Full Range); unit: kilograms per meter squared] | 30.17 [25.00 to 33.08] | 28.70 [26.98 to 30.42] | 29.68 [25.00 to 33.08]
History or Baseline Presence of Abnormality or Disease [Count of Participants; unit: Participants]
  Gastrointestinal | 4 | 2 | 6
  Head, Eyes, Ears, Nose, Throat | 4 | 2 | 6
  Musculoskeletal | 3 | 2 | 5
  Cardiovascular | 3 | 1 | 4
  Endocrine / Metabolic | 2 | 2 | 4
  Genitourinary | 4 | 0 | 4
  Respiratory | 4 | 0 | 4
  Dermatologic | 0 | 2 | 2
  Neurologic | 1 | 1 | 2
  Hematopoietic / Lymph | 1 | 0 | 1
  Neck | 1 | 0 | 1
  Breasts | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Proliferation Index (Ki-67) Expression, Assessed in Tumor Tissue by Immunohistochemistry
Description: Baseline, post-exposure, absolute change in Ki-67, and difference in absolute change between the ACTOplus met XR and placebo subjects will all be summarized with descriptive statistics. Ki-67 is a semi-quantitative immune-histochemistry analysis in which a computer generates an analysis based on the staining within tumor and normal cells leading to a score which is an indirect measure of cellular proliferation. Will compare the difference in absolute change in Ki-67 between the ACTOplus met XR and placebo arms using a two sided two-sample Student's t-test or Wilcoxon rank-sum test, as appropriate, at a significance level of 0.05.
Time Frame: Baseline to days 11-22
Population: 1 sample in the treatment group was not analyzed because site misplaced the sample.
Measure: Median (Inter-Quartile Range); unit: proliferation index expression
Arm/Group | Group I (ACTOplus Met XR) | Group II (Placebo)
Number analyzed (Participants) | 3 | 2
proliferation index expression
  baseline | 20.40 [19.84 to 25.10] | 13.69 [12.91 to 14.46]
  Day 11-22: number analyzed (Participants) | 3 | 1
  Day 11-22 | 17.57 [17.17 to 17.64] | 36.96 [36.96 to 36.96]
  absolute change from baseline: number analyzed (Participants) | 3 | 1
  absolute change from baseline | -2.68 [-7.46 to -2.60] | 24.82 [24.82 to 24.82]

2. Secondary Outcome: Change in Ki-67 Expression in Visually Normal Appearing Tissue, Assessed by Immunohistochemistry
Description: Will be summarized for baseline, post-exposure, and absolute change by treatment arm using the appropriate descriptive statistics, and will be evaluated with Student's t-test or Wilcoxon rank-sum test.
Time Frame: Baseline to days 11-22
Population: 1 sample in the treatment group was not analyzed because site misplaced the sample.
Measure: Median (Inter-Quartile Range); unit: proliferation index expression
Arm/Group | Group I (ACTOplus Met XR) | Group II (Placebo)
Number analyzed (Participants) | 3 | 2
proliferation index expression
  baseline | 17.58 [15.18 to 17.68] | 14.52 [11.66 to 17.38]
  Day 11-22: number analyzed (Participants) | 3 | 1
  Day 11-22 | 11.81 [10.02 to 14.23] | 26.05 [26.05 to 26.05]
  absolute change from baseline: number analyzed (Participants) | 3 | 1
  absolute change from baseline | -5.77 [-7.66 to -0.95] | 17.25 [17.25 to 17.25]

3. Secondary Outcome: Change in Cleaved Caspase 3 Expression in Visually Normal Appearing Tissue and Tumor Tissue Samples, Assessed by Immunohistochemistry
Description: Cleaved Caspase 3 is a semi-quantitative immune-histochemistry analysis in which a computer generates an analysis based on the staining within tumor and normal cells leading to a score which is a direct measure of cellular apoptosis. Will be summarized for baseline, post-exposure, and absolute change by treatment arm using the appropriate descriptive statistics, and will be evaluated with Student's t-test or Wilcoxon rank-sum test.
Time Frame: Baseline to days 11-22
Population: 1 sample in the treatment group was not analyzed because site misplaced the sample.
Measure: Mean (Standard Deviation); unit: percent positive cells
Arm/Group | Group I (ACTOplus Met XR) | Group II (Placebo)
Number analyzed (Participants) | 3 | 2
percent positive cells
  Baseline Tumor Tissue | 1.000 (1.000) | 1.000 (0.000)
  Post-Exposure Tumor Tissue: number analyzed (Participants) | 3 | 1
  Post-Exposure Tumor Tissue | 3.333 (4.041) | 4.000 (NA) — only 1 participant measured
  Baseline Normal Tissue | 0.000 (0.000) | 0.000 (0.000)
  Post-Exposure Normal Tissue: number analyzed (Participants) | 2 | 1
  Post-Exposure Normal Tissue | 0.000 (0.000) | 0.000 (NA) — only 1 participant measured

4. Secondary Outcome: Change in Cyclin D1, p21 and Biguanide or Phosphorylated AKT, Phosphorylated AMPK, Phosphorylated S6 (Metformin), and PPAR Gamma Expression, Assessed by Immunohistochemistry
Description: as for outcome 2
Time Frame: Baseline to days 11-22
Population: 1 sample in the treatment group was not analyzed because site misplaced the sample.
Measure: Median (Inter-Quartile Range); unit: percent positive cells
Arm/Group | Group I (ACTOplus Met XR) | Group II (Placebo)
Number analyzed (Participants) | 3 | 2
percent positive cells
  Cyclin D1 Baseline: number analyzed (Participants) | 2 | 2
  Cyclin D1 Baseline | 0.051 [0.039 to 0.062] | 0.020 [0.014 to 0.025]
  Cyclin D1 Day 11-22: number analyzed (Participants) | 3 | 1
  Cyclin D1 Day 11-22 | 0.050 [0.044 to 0.086] | 0.033 [0.033 to 0.033]
  Absolute change in Cyclin D1 from Baseline: number analyzed (Participants) | 2 | 1
  Absolute change in Cyclin D1 from Baseline | -0.0066 [-0.0210 to 0.0079] | 0.0019 [0.0019 to 0.0019]
  P21 Baseline: number analyzed (Participants) | 3 | 1
  P21 Baseline | 0.090 [0.077 to 0.166] | 0.112 [0.112 to 0.112]
  P21 Day 11-22: number analyzed (Participants) | 2 | 1
  P21 Day 11-22 | 0.068 [0.066 to 0.070] | 0.052 [0.052 to 0.052]
  Absolute change in P21 from Baseline: number analyzed (Participants) | 2 | 1
  Absolute change in P21 from Baseline | -0.0093 [-0.014 to -0.0049] | -0.0605 [-0.0605 to -0.0605]
  Phosphorylated AKT Baseline | 0.00018 [0.00015 to 0.00442] | 0.00013 [0.000067 to 0.00020]
  Phosphorylated AKT Day 11-22: number analyzed (Participants) | 3 | 1
  Phosphorylated AKT Day 11-22 | 0.00048 [0.00025 to 0.00481] | 0.00042 [0.00042 to 0.00042]
  Absolute change in phosphorylated AKT from baseline: number analyzed (Participants) | 2 | 1
  Absolute change in phosphorylated AKT from baseline | 0.00031 [0.00010 to 0.00039] | 0.00016 [0.00016 to 0.00016]
  Phosphorylated AMPK at Baseline: number analyzed (Participants) | 3 | 1
  Phosphorylated AMPK at Baseline | 0.079 [0.075 to 0.088] | 0.363 [0.363 to 0.363]
  Phosphorylated AMPK Day 11-22: number analyzed (Participants) | 3 | 1
  Phosphorylated AMPK Day 11-22 | 0.131 [0.103 to 0.134] | 0.030 [0.030 to 0.030]
  Absolute change in phosphorylated AMPK from baseline: number analyzed (Participants) | 3 | 1
  Absolute change in phosphorylated AMPK from baseline | 0.052 [0.015 to 0.06] | -0.333 [-0.333 to -0.333]
  PPAR gamma at Baseline | 0.0547 [0.0286 to 0.066] | 0.0138 [0.0072 to 0.020]
  PPAR gamma Day 11-22: number analyzed (Participants) | 3 | 1
  PPAR gamma Day 11-22 | 0.0061 [0.0056 to 0.020] | 0.0200 [0.0200 to 0.0200]
  Absolute change in PPAR gamma from baseline: number analyzed (Participants) | 3 | 1
  Absolute change in PPAR gamma from baseline | -0.022 [-0.047 to -0.0091] | 0.019 [0.019 to 0.0194]
  Phosphorylated S6 at Baseline | 0.284 [0.188 to 0.339] | 0.188 [0.143 to 0.232]
  Phosphorylated S6 Day 11-22: number analyzed (Participants) | 3 | 1
  Phosphorylated S6 Day 11-22 | 0.282 [0.226 to 0.298] | 0.071 [0.071 to 0.071]
  Absolute change in phosphorylated S6 from Baseline: number analyzed (Participants) | 3 | 1
  Absolute change in phosphorylated S6 from Baseline | 0.029 [-0.098 to 0.110] | -0.028 [-0.028 to -0.028]

5. Secondary Outcome: Change in Regulatory T Cell, T4, T8, Tumor-associated Macrophage-CD68 Positive, PD1, PD-L1 Expression, Assessed in Tumor Tissue by Immunohistochemistry
Description: as for outcome 2
Time Frame: Baseline to days 11-22
Population: 1 sample in the treatment group was not analyzed because site misplaced the sample.
Measure: Median (Inter-Quartile Range); unit: percent positive cells
Arm/Group | Group I (ACTOplus Met XR) | Group II (Placebo)
Number analyzed (Participants) | 3 | 2
percent positive cells
  CD68 Baseline: number analyzed (Participants) | 2 | 2
  CD68 Baseline | 0.11 [0.070 to 0.14] | 0.190 [0.175 to 0.21]
  CD68 Day 11-22: number analyzed (Participants) | 3 | 1
  CD68 Day 11-22 | 0.10 [0.074 to 0.11] | 0.23 [0.227 to 0.23]
  Absolute Change in CD68 from Baseline: number analyzed (Participants) | 2 | 1
  Absolute Change in CD68 from Baseline | -0.033 [-0.055 to -0.010] | 0.068 [0.068 to 0.068]
  PD1 Baseline | 0.0520 [0.0439 to 0.153] | 0.0356 [0.0290 to 0.042]
  PD1 Day 11-22: number analyzed (Participants) | 3 | 1
  PD1 Day 11-22 | 0.0088 [0.0081 to 0.017] | 0.0721 [0.0721 to 0.0721]
  Absolute Change in PD1 from Baseline: number analyzed (Participants) | 3 | 1
  Absolute Change in PD1 from Baseline | -0.045 [-0.15 to -0.027] | 0.050 [0.05 to 0.050]
  PD-L1 Baseline: number analyzed (Participants) | 2 | 2
  PD-L1 Baseline | 0.0632 [0.0335 to 0.093] | 0.0086 [0.0051 to 0.012]
  PD-L1 Day 11-22: number analyzed (Participants) | 3 | 1
  PD-L1 Day 11-22 | 0.0494 [0.0263 to 0.051] | 0.0136 [0.0136 to 0.0136]
  Absolute Change in PD-L1 from Baseline: number analyzed (Participants) | 2 | 1
  Absolute Change in PD-L1 from Baseline | -0.012 [-0.043 to 0.019] | 0.012 [0.012 to 0.012]
  CD8 Baseline: number analyzed (Participants) | 2 | 2
  CD8 Baseline | 0.244 [0.180 to 0.31] | 0.141 [0.122 to 0.16]
  CD8 Day 11-22: number analyzed (Participants) | 2 | 1
  CD8 Day 11-22 | 0.095 [0.066 to 0.12] | 0.189 [0.189 to 0.19]
  Absolute Change in CD8 from Baseline: number analyzed (Participants) | 1 | 1
  Absolute Change in CD8 from Baseline | -0.218 [-0.218 to -0.218] | 0.086 [0.086 to 0.086]
  CD4 Baseline | 0.193 [0.114 to 0.204] | 0.195 [0.191 to 0.198]
  CD4 Day 11-22: number analyzed (Participants) | 3 | 1
  CD4 Day 11-22 | 0.159 [0.118 to 0.332] | 0.074 [0.074 to 0.074]
  Absolute Change in CD4 from Baseline: number analyzed (Participants) | 3 | 1
  Absolute Change in CD4 from Baseline | 0.043 [-0.0064 to 0.18] | -0.128 [-0.128 to -0.128]
  FoxP3 Baseline | 0.027 [0.015 to 0.035] | 0.057 [0.036 to 0.079]
  FoxP3 Day 11-22: number analyzed (Participants) | 3 | 1
  FoxP3 Day 11-22 | 0.020 [0.014 to 0.025] | 0.038 [0.038 to 0.038]
  Absolute Change in FoxP3 from Baseline: number analyzed (Participants) | 2 | 1
  Absolute Change in FoxP3 from Baseline | 0.0034 [-0.010 to 0.0041] | 0.0235 [0.0235 to 0.0235]

6. Secondary Outcome: Genes With Significant Changes From Baseline to Days 11-22 in Tumor Tissue in Treated Participants: Change in Whole Transcriptome Gene Analysis on Total Ribonucleic Acid Samples
Description: as for outcome 2
Time Frame: Baseline to days 11-22
Population: Pre- and post-treatment RNA-seq data was available in four ACTOplus treated participants and one placebo treated participant. Because of this, a comparison between the treatment arms was not deemed to be possible or useful. What was attempted was an analysis of change from baseline values for the ACTOplus met® XR arm.
Measure: Mean (Standard Deviation); unit: raw counts of RNA sequencing reads
Units Other Than Participants: genes
Groups:
- Group I ACTOplus Met XR: Patients receive ACTOplus met XR PO QD for 10-21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Group I ACTOplus Met XR | Group II (Placebo)
Number analyzed (Participants) | 4 | 1
Number analyzed (genes) | 37769 | 37769
raw counts of RNA sequencing reads
  ENSG00000229822: number analyzed (genes) | 1 | 1
  ENSG00000229822 | 1.0011 (0.0240) | -5.0023 (NA) — only 1 data point
  ENSG00000230585: number analyzed (genes) | 1 | 1
  ENSG00000230585 | -1.0217 (0.0257) | -3.0108 (NA) — only 1 data point
  ENSG00000249245: number analyzed (genes) | 1 | 1
  ENSG00000249245 | -1.0098 (0.0050) | 0.0000 (NA) — only 1 data point
  ENSG00000261792: number analyzed (genes) | 1 | 1
  ENSG00000261792 | 1.0007 (0.0063) | 0.0000 (NA) — only 1 data point
Statistical Analysis 1: Comparison: Group I ACTOplus Met XR; ENSG00000229822 baseline and post exposure; Test type: Superiority; p = 0.031, Benjamini and Hochberg; Mean Difference (Final Values) = 1.0011, Standard Deviation 0.0240
Statistical Analysis 2: Comparison: Group I ACTOplus Met XR; ENSG00000230585 baseline and post exposure; Test type: Superiority; p = 0.031, Benjamini and Hochberg; Mean Difference (Final Values) = -1.0217, Standard Deviation 0.0257
Statistical Analysis 3: Comparison: Group I ACTOplus Met XR; ENSG00000249245 baseline and post exposure; Test type: Superiority; p < 0.001, Benjamini and Hochberg; Mean Difference (Final Values) = -1.0098, Standard Deviation 0.0050
Statistical Analysis 4: Comparison: Group I ACTOplus Met XR; ENSG00000261792 baseline and post exposure; Test type: Superiority; p < 0.001, Benjamini and Hochberg; Mean Difference (Final Values) = 1.0007, Standard Deviation 0.0063

7. Secondary Outcome: Genes With Significant Changes From Baseline to Days 11-22 for Normal Tissue: Change in Whole Transcriptome Gene Analysis on Total Ribonucleic Acid Samples
Description: as for outcome 2
Time Frame: Baseline to days 11-22
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: raw counts of RNA sequencing reads
Units Other Than Participants: genes
Arm/Group | Group I ACTOplus Met XR | Group II (Placebo)
Number analyzed (Participants) | 4 | 1
Number analyzed (genes) | 1 | 1
raw counts of RNA sequencing reads | 1.0060 (0.0060) | 2.0135 (NA) — only 1 data point
Statistical Analysis 1: Comparison: Group I ACTOplus Met XR; ENSG00000234806 baseline and post exposure; Test type: Superiority; p = 0.002, Benjamini and Hochberg; Mean Difference (Final Values) = 1.0060, Standard Deviation 0.0060

8. Secondary Outcome: Genes With Significant Changes From Baseline to Days 11-22 for Tumor-Normal Tissue: Change in Whole Transcriptome Gene Analysis on Total Ribonucleic Acid Samples
Description: The plan was to summarize for baseline, post-exposure, and absolute change by treatment arm using the appropriate descriptive statistics, and will be evaluated with Student's t-test or Wilcoxon rank-sum test.
Time Frame: Baseline to days 11-22
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: raw counts of RNA sequencing reads
Units Other Than Participants: genes
Arm/Group | Group I ACTOplus Met XR | Group II (Placebo)
Number analyzed (Participants) | 4 | 1
Number analyzed (genes) | 37769 | 37769
raw counts of RNA sequencing reads
  ENSG00000232479: number analyzed (genes) | 1 | 1
  ENSG00000232479 | 1.0013 (0.0072) | -1.0087 (NA) — only 1 data point
  ENSG00000233163: number analyzed (genes) | 1 | 1
  ENSG00000233163 | 1.0037 (0.0193) | -1.0003 (NA) — only 1 data point
  ENSG00000249245: number analyzed (genes) | 1 | 1
  ENSG00000249245 | -1.0098 (0.0050) | 0.0000 (NA) — only 1 data point
Statistical Analysis 1: Comparison: Group I ACTOplus Met XR; ENSG00000232479 baseline and post exposure; Test type: Superiority; p = 0.002, Benjamini and Hochberg; Mean Difference (Final Values) = 1.0013, Standard Deviation 0.0072
Statistical Analysis 2: Comparison: Group I ACTOplus Met XR; ENSG00000233163 baseline and post exposure; Test type: Superiority; p = 0.020, Benjamini and Hochberg; Mean Difference (Final Values) = 1.0037, Standard Deviation 0.0193
Statistical Analysis 3: Comparison: Group I ACTOplus Met XR; ENSG00000249245 baseline and post-exposure; Test type: Superiority; p = 0.001, Benjamini and Hochberg; Mean Difference (Final Values) = -1.0098, Standard Deviation 0.0050

9. Secondary Outcome: Human Papillomavirus Status Assessed in Tumor Tissue by p16 by Immunohistochemistry
Description: Human papillomavirus status will be assessed in tumor tissue by p16 by immunohistochemistry.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (ACTOplus Met XR) | Group II (Placebo)
Number analyzed (Participants) | 4 | 2
Participants
  Positive | 2 | 0
  Not Tested | 2 | 2

10. Other Pre Specified Outcome: Change in Tumor Fluorodeoxyglucose Uptake/Metabolism Assess by Treatment Positron Emission Tomography/Computed Tomography
Description: Tumor fluorodeoxyglucose uptake/metabolism assess by treatment positron emission tomography/computed tomography.
Time Frame: Baseline to days 11-22
Population: No one consented to this aspect of the study, no data is available.
Arm/Group | Group I (ACTOplus Met XR) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 22 days
Arm/Group | Group I (ACTOplus Met XR) | Group II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (ACTOplus Met XR) (N=4) | Group II (Placebo) (N=2)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) — this adverse event was reported by the participant prior to randomization
Fatigue (General disorders) | 1 (1) | 0 (0) — this adverse event was reported by the participant prior to randomization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT02917629/Prot_SAP_000.pdf